CLINICAL TRIAL: NCT03293953
Title: Prospective Comparison Between Transient Elastography (TE), Shear Wave Elastography (SWE) and Magnetic Resonance Elastography (MRE) for Non-invasive Assessment of Liver Fibrosis in Patients Affected by Chronic Viral Hepatitis
Brief Title: Prospective Comparison Between TE, SWE and MRE (FULLFIBRO01)
Acronym: FULLFIBRO01
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ente Ospedaliero Ospedali Galliera (Other)
Collaborators: General Electric (Industry)
Responsible Party: Principal Investigator, Gian Andrea Rollandi, Direttore medico responsabile S.C. Radiodiagnostica, Ente Ospedaliero Ospedali Galliera
Other Study IDs: 41UCS2016
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Liver Fibrosis
Keywords: HCV; HIV; Liver Fibrosis; Liver Iron Overload
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of the present study is to compare the diagnostic performance of three non-invasive stiffness imaging methods (TE, SWE and MRE) in a consecutive cohort of patients with chronic viral C hepatitis or co-infected by HCV+ Human Human Immunodeficiency Virus (HIV).

DETAILED DESCRIPTION:
Primary Endpoint: Verify if Transient Elastography, Shear Wave Elastography, Magnetic Resonance Elastography (MRE) get comparable results in the measurement of liver fibrosis Secondary Endpoint: To evaluate if the level of liver iron overload and steatosis may act as a confounding factor in stiffness measurements by MRE.

Tertiary Endpoint: to provide information about the prevalence and grade of steatosis in a consecutive cohort of patients with chronic viral C hepatitis, and to verify if the presence and grade of parenchymal steatosis may affect the correlation between the different non-invasive stiffness imaging modalities.

Subject: consecutive 100 patients affected by chronic viral C hepatitis or co-infected by HCV+ Human Human Immunodeficiency Virus (HIV).

ELIGIBILITY:
Inclusion Criteria:

* enrollment of a consecutive cohort of at least 100 patients affected by chronic C virus hepatitis (HCV) or co-infected by HCV+ Human Immunodeficiency Virus (HIV).

Exclusion Criteria:

* contraindications to undergo MRI examination. Impossibility to obtain a valid TE measurement (e.g. narrow intercostal spaces; obese patients)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients affected by chronic C virus hepatitis (HCV) or co-infected by HCV+ Human Immunodeficiency Virus (HIV)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
liver stiffness | 18 months
  liver stiffness is indicated in kPa

SECONDARY OUTCOMES:
liver iron overload | 18 months
  liver iron concentration (LIC) is indicated in mg/g dw
liver steatosis | 18 months
  liver steatosis

CONTACTS AND LOCATIONS:
Overall Officials: Gian Andrea Rollandi, MD, Principal Investigator — Direttore SC Radiodiagnostica, Coordinatore Scientifico EO Ospedali Galliera Genova-Italy
Locations (1):
- SC Radiodiagnostica, Genova, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ghany MG, Strader DB, Thomas DL, Seeff LB; American Association for the Study of Liver Diseases. Diagnosis, management, and treatment of hepatitis C: an update. Hepatology. 2009 Apr;49(4):1335-74. doi: 10.1002/hep.22759. No abstract available. PMID 19330875
- [Background] Castera L. Invasive and non-invasive methods for the assessment of fibrosis and disease progression in chronic liver disease. Best Pract Res Clin Gastroenterol. 2011 Apr;25(2):291-303. doi: 10.1016/j.bpg.2011.02.003. PMID 21497746
- [Background] Bravo AA, Sheth SG, Chopra S. Liver biopsy. N Engl J Med. 2001 Feb 15;344(7):495-500. doi: 10.1056/NEJM200102153440706. No abstract available. PMID 11172192
- [Background] Regev A, Berho M, Jeffers LJ, Milikowski C, Molina EG, Pyrsopoulos NT, Feng ZZ, Reddy KR, Schiff ER. Sampling error and intraobserver variation in liver biopsy in patients with chronic HCV infection. Am J Gastroenterol. 2002 Oct;97(10):2614-8. doi: 10.1111/j.1572-0241.2002.06038.x. PMID 12385448
- [Background] Baranova A, Lal P, Birerdinc A, Younossi ZM. Non-invasive markers for hepatic fibrosis. BMC Gastroenterol. 2011 Aug 17;11:91. doi: 10.1186/1471-230X-11-91. PMID 21849046
- [Background] Paparo F, Corradi F, Cevasco L, Revelli M, Marziano A, Molini L, Cenderello G, Cassola G, Rollandi GA. Real-time elastography in the assessment of liver fibrosis: a review of qualitative and semi-quantitative methods for elastogram analysis. Ultrasound Med Biol. 2014 Sep;40(9):1923-33. doi: 10.1016/j.ultrasmedbio.2014.03.021. Epub 2014 Jun 25. PMID 24972497
- [Background] Tang A, Cloutier G, Szeverenyi NM, Sirlin CB. Ultrasound Elastography and MR Elastography for Assessing Liver Fibrosis: Part 1, Principles and Techniques. AJR Am J Roentgenol. 2015 Jul;205(1):22-32. doi: 10.2214/AJR.15.14552. Epub 2015 Apr 23. PMID 25905647
- [Background] Ferraioli G, Tinelli C, Lissandrin R, Zicchetti M, Dal Bello B, Filice G, Filice C. Point shear wave elastography method for assessing liver stiffness. World J Gastroenterol. 2014 Apr 28;20(16):4787-96. doi: 10.3748/wjg.v20.i16.4787. PMID 24782633
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: management of hepatitis C virus infection. J Hepatol. 2011 Aug;55(2):245-64. doi: 10.1016/j.jhep.2011.02.023. Epub 2011 Mar 1. No abstract available. PMID 21371579
- [Background] Tang A, Cloutier G, Szeverenyi NM, Sirlin CB. Ultrasound Elastography and MR Elastography for Assessing Liver Fibrosis: Part 2, Diagnostic Performance, Confounders, and Future Directions. AJR Am J Roentgenol. 2015 Jul;205(1):33-40. doi: 10.2214/AJR.15.14553. Epub 2015 Apr 23. PMID 25905762
- [Background] Ziol M, Handra-Luca A, Kettaneh A, Christidis C, Mal F, Kazemi F, de Ledinghen V, Marcellin P, Dhumeaux D, Trinchet JC, Beaugrand M. Noninvasive assessment of liver fibrosis by measurement of stiffness in patients with chronic hepatitis C. Hepatology. 2005 Jan;41(1):48-54. doi: 10.1002/hep.20506. PMID 15690481
- [Background] Yoon JH, Lee JM, Joo I, Lee ES, Sohn JY, Jang SK, Lee KB, Han JK, Choi BI. Hepatic fibrosis: prospective comparison of MR elastography and US shear-wave elastography for evaluation. Radiology. 2014 Dec;273(3):772-82. doi: 10.1148/radiol.14132000. Epub 2014 Jul 7. PMID 25007047
- [Background] Bohte AE, de Niet A, Jansen L, Bipat S, Nederveen AJ, Verheij J, Terpstra V, Sinkus R, van Nieuwkerk KM, de Knegt RJ, Baak BC, Jansen PL, Reesink HW, Stoker J. Non-invasive evaluation of liver fibrosis: a comparison of ultrasound-based transient elastography and MR elastography in patients with viral hepatitis B and C. Eur Radiol. 2014 Mar;24(3):638-48. doi: 10.1007/s00330-013-3046-0. Epub 2013 Oct 25. PMID 24158528
- [Background] Paparo F, Cenderello G, Revelli M, Bacigalupo L, Rutigliani M, Zefiro D, Cevasco L, Amico M, Bandelloni R, Cassola G, Forni GL, Rollandi GA. Diagnostic value of MRI proton density fat fraction for assessing liver steatosis in chronic viral C hepatitis. Biomed Res Int. 2015;2015:758164. doi: 10.1155/2015/758164. Epub 2015 Mar 19. PMID 25866807
- [Background] Negro F. Mechanisms and significance of liver steatosis in hepatitis C virus infection. World J Gastroenterol. 2006 Nov 14;12(42):6756-65. doi: 10.3748/wjg.v12.i42.6756. PMID 17106922
- [Background] Sun HY, Lee JM, Han JK, Choi BI. Usefulness of MR elastography for predicting esophageal varices in cirrhotic patients. J Magn Reson Imaging. 2014 Mar;39(3):559-66. doi: 10.1002/jmri.24186. Epub 2013 Sep 23. PMID 24115368
- [Background] Manduca A, Oliphant TE, Dresner MA, Mahowald JL, Kruse SA, Amromin E, Felmlee JP, Greenleaf JF, Ehman RL. Magnetic resonance elastography: non-invasive mapping of tissue elasticity. Med Image Anal. 2001 Dec;5(4):237-54. doi: 10.1016/s1361-8415(00)00039-6. PMID 11731304
- [Background] Bydder M, Yokoo T, Hamilton G, Middleton MS, Chavez AD, Schwimmer JB, Lavine JE, Sirlin CB. Relaxation effects in the quantification of fat using gradient echo imaging. Magn Reson Imaging. 2008 Apr;26(3):347-59. doi: 10.1016/j.mri.2007.08.012. Epub 2008 Feb 21. PMID 18093781
- [Background] Angelucci E, Giovagnoni A, Valeri G, Paci E, Ripalti M, Muretto P, McLaren C, Brittenham GM, Lucarelli G. Limitations of magnetic resonance imaging in measurement of hepatic iron. Blood. 1997 Dec 15;90(12):4736-42. PMID 9389689
- [Background] Paparo F, Cevasco L, Zefiro D, Biscaldi E, Bacigalupo L, Balocco M, Pongiglione M, Banderali S, Forni GL, Rollandi GA. Diagnostic value of real-time elastography in the assessment of hepatic fibrosis in patients with liver iron overload. Eur J Radiol. 2013 Dec;82(12):e755-61. doi: 10.1016/j.ejrad.2013.08.038. Epub 2013 Aug 30. PMID 24050879